CLINICAL TRIAL: NCT00866385
Title: An Open, Randomised, Phase I, 2-Period Crossover Trial to Investigate the Absolute Bioavailability and the Effect of Food on the Oral Bioavailability of AZD8566 in Healthy Volunteers
Brief Title: AZD8566 Food Effect/Microtracer Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: H Parmar MD, (Acting) Medical Science Director, Respiratory and, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D1320C00011; Pharmaceutical Profiles PL1168
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2009-06-09 (Estimated); Status verified 2009-06

CONDITIONS: Healthy Volunteer Study
Keywords: Healthy Volunteer; AZD8566; Food Effect; Microtracer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AZD8566 — Single 6 mg oral solution dose
Drug: AZD8566 IV carbon labelled — Single 10 mcg intravenous carbon-14 microtracer dose

SUMMARY:
A study designed to look at how the drug AZD8566 is taken up by the body when given with or without food. In some subjects a comparison will be made with a very small labelled microdose given into a vein.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Clinically normal physical findings and laboratory values as judged by the investigator with normal ECG
* Females who are permanently or surgically sterile or post-menopausal and males

Exclusion Criteria:

* History of any convulsions or seizures
* History of infection or risk of infection due to recent surgery or trauma
* History or presence of conditions know to interfere with the absorption, distribution, metabolism and excretion of the study drug

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2009-03; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile: concentration of AZD8566 in blood in the presence or absence of food | Samples taken during visit 2 and visit 3, at up to 16 defined timepoints pre and post dose

SECONDARY OUTCOMES:
Safety and tolerability of AZD8566 in healthy volunteers in the fed and fasted state by assessment of vital signs, laboratory variables, ECGs and adverse events | Assessments taken during visit 1 and at defined timepoints pre and post dose during visits 2 and 3. Volunteers will be monitored throughout the study for adverse events.
Bioavailability of an oral solution formulation of AZD8566 in the fasted state compared with an intravenous carbon-14 microtracer dose | Samples taken during visit 2, at up to 40 defined timepoints pre and post dose
Intravenous pharmacokinetics | Samples taken during visit 2, at up to 40 defined timepoints pre and post dose

CONTACTS AND LOCATIONS:
Overall Officials: Jo Collier, Dr,MB, ChB, Principal Investigator — Pharmaceutical Profiles, Mere Way, Ruddington Fields, Nottingham NG11 6JS
Locations (1):
- Research Site, Nottingham, United Kingdom